CLINICAL TRIAL: NCT04118647
Title: Effective Mechanisms of Wu-Chu-Yu Tang on Gastroesophageal Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH108-REC2-101
Record Dates: First submitted 2019-09-18; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Wu-Chu-Yu Tang; Gastroesophageal Reflux Disorder; 24 Hours Esophageal PH and Multichannel Intraluminal Impedance Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wu-Chu-Yu tang (Experimental)
  Interventions: Drug: Wu-Chu-Yu tang

INTERVENTIONS:
Drug: Wu-Chu-Yu tang — Wu-Chu-Yu tang at a rate of 3.0 g three times per day for 28 days.

SUMMARY:
Gastroesophageal reflux disorder (GERD) is due to gastric content reflux to esophagus cause symptom and complication including intra-esophagus such as reflux esophagitis, and extra-esophagus such as cough etc. Because the changes of dietary habit, and improvement of examination skill and data analysis, the prevalence of GERD increased 2.5 multiple from 1995 to 2002, and suggesting the prevalence is 25% in Taiwan community.

The etiology of GERD is multi-effect, such as transient lower esophageal sphincter relaxation and abnormal pressure of lower esophageal sphincter, which may induced the esophageal mucosal injury by gastric acid, bile or pancreases enzyme.

Wu-Chu-Yu tang consists of Evodia fargesii Dode (Evodia Fruit), Panax ginseng C. (Ginseng), Ziziphus jujube Mill (Chinses Date), Zingiber officinale Rosee (Fresh Ginger).According to "I-Fang-Chi-Chieh" and "Shanghonzobinglun" recordings that Wu-Chu-Yu tang can treat vomiting, and also can relax gastric tonicity and can enhance peristalsis of stomach. According to Randomized, double blind, placebo control trial to evaluate the efficacy of Wu-Chu-Yu Tang on gastroesophageal reflux disease, we know the Wu-Chu-Yu tang have the equivalent effect proton pump inhibitor omeprazole. But, the mechanism of Wu-Chu-Yu tang is still unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Gender：male or female.
2. Age：from 20 years old (inclusive) to 75 years old (inclusive).
3. Diagnosis of gastroesophageal reflux disease.
4. there is a heartburn or acid regurgitation phenomenon.
5. After detailed description of the entire research purpose or process, voluntarily participate in the study and sign the consent form.

Exclusion Criteria:

1. Exclude peptic ulcers, gallstones (including intrahepatic and common bile ducts) and major diseases such as: cancer, congestive hear failured NYHA class>II, COPD attack.
2. Barrett's esophagus, narrow esophagus or caustic injury of upper gastrointestinal tract.
3. History of esophagus and gastroduodenal surgery.
4. Tarry stool suspected gastrointestinal bleeding.
5. History of alcohol or drug abuse.
6. Patients with a history of allergies to the test drug.
7. Can not cooperate with mental illness.
8. Pregnant women or women who are breastfeeding.
9. Liver function SGOT and SGPT are more than twice the normal value.
10. renal function test BUN, Creatinine is greater than the normal value.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
24 hours esophageal PH | 28 days
  Analysis the 24 hours PH change
DeMeester score | 28 days
  DeMeester score had two major component as 1.total time of pH<4(%) and 2.number of reflux episode. Each major part had two minor component.Fist one, percentage of total time pH<4, had 1. percentage of upright time when pH<4 and 2.percentage of supine time when pH<4. Secondary part, number of reflux episode, had 1.number of reflux episode over 5 mintues and 2.longest reflux time. Finally, there was a composite score as the DeMeester score.

SECONDARY OUTCOMES:
Reflux Disease Questionnaire | 56 days
  Reflux Disease Questionnaire had one major component as Thinking about your symptoms over the past 7 days, how often have you had the following? And then there were six minor component: a. A burning feeling behind your breastbone b. Pain behind your breastbone c. A burning feeling in the centre of the upper stomach d. Pain in the centre of the upper stomach e. An acid taste in your mouth f. Unpleasant movement ofmaterial upwards from the stomach. Each question was different frequency as have not had, 1 day, 2 days, 3-4 days, 5-6 days or daily in one week.
  Each frequency had one score and subscale had score from one to six. The total score was one to thirty six. The score more less means more better outcome.
SF-36 questionnaire | 56 days
  The scores of each question are added together to obtain the scale. The total score, the higher the total score, the quality of healthy life The higher.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided